CLINICAL TRIAL: NCT07033273
Title: The Predictive Value of the Inferior Vena Cava Collapsibility Index for Intradialytic Hypotension: A Prospective Multicenter Observational Stud
Brief Title: Inferior Vena Cava Collapsibility Index and Intradialytic Hypotension
Acronym: IVC-HD
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Wuhu County Traditional Chinese Medicine Hospital (Other); Wuhu City Second People's Hospital (Other)
Responsible Party: Principal Investigator, Qiancheng Xu, Principal Investigator, First Affiliated Hospital of Wannan Medical College
Other Study IDs: 2025-37
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: End-Stage Renal Disease Requiring Haemodialysis; Intradialytic Hypotension
Keywords: Intradialytic Hypotension; Hemodialysis; Inferior Vena Cava Collapsibility Index; Blood Pressure Prediction; Vascular Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maintenance Hemodialysis Patients: Adult patients with end-stage renal disease undergoing maintenance hemodialysis for at least three months, assessed for intradialytic hypotension risk using ultrasound measurements of the Inferior Vena Cava Collapsibility Index (IVCCI).
  Interventions: Other: Non-invasive Monitoring

INTERVENTIONS:
Other: Non-invasive Monitoring — All participants will undergo non-invasive measurement of Inferior Vena Cava Collapsibility Index (IVCCI) using ultrasound and routine blood pressure monitoring before and during hemodialysis sessions. No treatment or experimental intervention will be applied.

SUMMARY:
This multicenter, prospective observational study aims to evaluate the predictive value of the Inferior Vena Cava Collapsibility Index (IVCCI), along with IVC maximum diameter (IVCmax) and IVC minimum diameter (IVCmin), for intradialytic hypotension in patients undergoing maintenance hemodialysis. The study will be conducted at The First Affiliated Hospital of Wannan Medical College, Wuhu City Second People's Hospital, Wuhu Hospital of Chinese Traditional Medicine, Wuhu Jinghu District Hospital, and Wuhu Guangji Hospital. Eligible participants are adults aged 18 years or older with diagnosed end-stage renal disease (ESRD), receiving regular hemodialysis for at least three months. Patients with acute kidney injury, severe cardiac conditions, or other factors likely to influence results will be excluded.

Ultrasound measurements of IVCCI, IVCmax, and IVCmin will be performed once, precisely at 1 hour after dialysis initiation. IVCmax will be measured during inspiration when the IVC is at its largest, and IVCmin during expiration when it is at its smallest. Blood pressure will be monitored continuously during the procedure. The primary objective is to assess the sensitivity, specificity, and optimal cutoff values of IVCCI, IVCmax, and IVCmin for predicting hypotension, aiming to provide a simple and non-invasive tool to facilitate personalized dialysis management and reduce intradialytic hypotension. A sample size of 188 participants is estimated, with data analyzed using ROC curves and multivariate regression methods. The study protocol adheres to ethical standards and regulatory requirements, demonstrating potential to improve patient safety and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with end-stage renal disease (ESRD).
* Undergoing regular hemodialysis for at least three months.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Hemodynamically unstable patients or those requiring vasopressor support.
* Patients with severe cardiac conditions, including congestive heart failure -classified as NYHA Class III-IV or severe valvular disease.
* Patients with known allergies to dialysis filters.
* Dialysis sessions terminated for reasons unrelated to hypotension (e.g., technical issues, patient request).
* Patients who withdraw informed consent during the study.
* Use of antihypertensive medications during dialysis sessions.
* Inability to undergo ultrasound assessment due to factors such as severe obesity or wounds obstructing access.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 80 years with end-stage renal disease who have been receiving maintenance hemodialysis for more than three months at participating dialysis centers. Participants are required to be able to provide informed consent and cooperate with study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of IVCCI at 1 Hour for Intradialytic Hypotension | 1 hour after dialysis initiation
  The IVC diameters willbe measured using bedside ultrasonography with a portable ultrasound device. The probe will be placed subcutaneously on the right side of the abdomen, along the mid-axillary line, approximately 2-3 cm below the hepatic vein confluence.End-expiratory diameter (IVCmin): measured during expiration when the IVC is at its smallest. End-inspiratory diameter (IVCmax): measured during inspiration when the IVC is at its largest.
  IVCCI calculated as (IVCmin-IVCmax)/IVCmax × 100% measured 1 hour after dialysis initiation.The sensitivity, specificity, and area under the ROC curve of dIVC in predicting hypotension events during dialysis.
Predictive Value of IVCmax at 1 Hour for Intradialytic Hypotension | 1 hour after dialysis initiation
  The sensitivity, specificity, and ROC of IVCmax measured 1 hour after dialysis initiation in predicting hypotension.
Predictive Value of IVCmin at 1 Hour for Intradialytic Hypotension | 1 hour after dialysis initiation.
  The sensitivity, specificity, and ROC of IVCmin measured 1 hour after dialysis initiation in predicting hypotension.

SECONDARY OUTCOMES:
Incidence of Intradialytic Hypotension | Up to one dialysis session (4 hours)
  The proportion of dialysis sessions experiencing hypotension, defined as a systolic blood pressure decrease ≥20 mmHg or associated symptoms.
Correlation Between IVC Parameters and Blood Pressure Changes | Up to one dialysis session (4 hours)
  Analysis of the correlation between IVCmax, IVCmin, and IVCCI measured at 1 hour and changes in systolic, diastolic, and mean arterial pressure from start to 1 hour.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wannan Medical College (Yijishan Hospital of Wannan Medical College), Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: No